CLINICAL TRIAL: NCT01969799
Title: A Randomized Blinded, Placebo-Controlled, Phase 2 Study of Aerosolized Amikacin and Fosfomycin Delivered Via the Investigational eFlow® Inline System in Mechanically Ventilated Patients With Gram-negative Bacterial Pneumonia (IASIS)
Brief Title: Aerosolized Amikacin and Fosfomycin in Mechanically Ventilated Patients With Gram-negative Pneumonia
Acronym: IASIS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cardeas Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAP-01-102; 2013-002855-13 (EudraCT Number)
Record Dates: First submitted 2013-10-22; First posted 2013-10-25 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2016-03

CONDITIONS: Pneumonia, Bacterial
Keywords: Gram-negative pneumonia; Aerosol antibiotics; Mechanical ventilation; Amikacin; Fosfomycin; Pneumonia, Bacterial; Pneumonia; Bacterial Infections; Lung Diseases; Respiratory Tract Diseases; Respiratory Tract Infections; Anti-Bacterial Agents; Anti-Infective Agents; Therapeutic Uses; Pharmacologic Actions
MeSH Terms: conditions — Pneumonia, Bacterial; Pneumonia; Bacterial Infections; Lung Diseases; Respiratory Tract Diseases; Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Amikacin fosfomycin inhalation solution (Experimental): 300 mg of amikacin and 120 mg of fosfomycin twice daily for 10 days to be administered by aerosol via the eFlow Inline System.
  Interventions: Drug: Amikacin fosfomycin inhalation solution
- Aerosolized placebo (Placebo Comparator): Aerosolized placebo twice daily for 10 days administered using the eFlow Inline System
  Interventions: Drug: Aerosolized placebo

INTERVENTIONS:
Drug: Amikacin fosfomycin inhalation solution — 300 mg of amikacin and 120 mg of fosfomycin twice daily for 10 days to be administered by aerosol via the eFlow Inline System
  Other Names: Amikacin fosfomycin inhalation system (AFIS); eFlow Inline System
  Arms: Amikacin fosfomycin inhalation solution
Drug: Aerosolized placebo — Placebo twice daily for 10 days to be administered by aerosol the eFlow Inline System
  Other Names: eFlow Inline System
  Arms: Aerosolized placebo

SUMMARY:
To demonstrate the safety and efficacy of adjunctive therapy with the Amikacin fosfomycin inhalation system (AFIS) versus aerosolized placebo to treat Gram-negative pneumonia in mechanically ventilated patients receiving IV antibiotics.

DETAILED DESCRIPTION:
The primary purpose of this study is to demonstrate the safety and efficacy of the amikacin fosfomycin inhalation system (AFIS). AFIS consists of amikacin solution and fosfomycin solution, delivered by aerosol to the lungs via the PARI Investigational eFlow Inline System (eFlow Inline System). All patients will receive a standardized course of intravenous (IV) antibiotics for a minimum of 7 days. Patients will be randomized to receive 10 days of treatment with either AFIS or placebo, in addition to the IV therapy. The primary efficacy endpoint is defined as the change from baseline in the Clinical Pulmonary Infection Score (CPIS) during the randomized course of study drug. The study was designed to enroll up to 150 patients with the desire to enroll at least 140 patients with gram negative pneumonia. The study was terminated at 143 when that goal was achieved

ELIGIBILITY:
Inclusion Criteria:

* Males and non-pregnant, non-lactating females, ≥ 18 years and ≤ 80 years of age
* Intubated and mechanically ventilated
* Diagnosis of pneumonia, defined as presence of a new or progressive infiltrate(s) on the most recent chest radiograph prior to screening, as determined by the treating physician
* Signs of infection (within 24 hours prior to screening):

  1. Fever (> 38ºC or > 100.4ºF); or
  2. Leukopenia (< 4,000 WBC/mm3) or leukocytosis (≥ 12,000 WBC/mm3)
* Impaired oxygenation (within 24 hours prior to screening):

  a. PaO2/FiO2 ≤ 350 mmHg
* Acute Physiology and Chronic Health Evaluation (APACHE) II score > 10 (within 24 hours prior to screening)
* Presence, or high suspicion, of Gram-negative organism(s) by either Gram stain or culture of respiratory secretions from a sample obtained within the previous 7 days (enrollment can occur before culture results are available)

Exclusion Criteria:

* History of hypersensitivity to amikacin, other aminoglycosides, fosfomycin, imipenem, meropenem, or colistin
* Received systemic antibiotic therapy for this episode of Gram-negative pneumonia for greater than 72 hours at the time of randomization
* PaO2/FiO2 ≤ 100 mmHg and diffuse infiltrates on Chest X-ray
* Refractory septic shock (severe sepsis plus unstable hypotension, in spite of adequate fluid resuscitation and vasopressors)
* Any of the following conditions that interfere with the assessment or interpretation of the diagnosis or response to therapy:

  1. chest trauma with ongoing loss of stability of the thoracic cage following a fracture of the sternum, ribs, or both;
  2. increased amounts of fluid in the lung cavities requiring chest tube drainage;
  3. lung cancer within the last 2 years;
  4. lung abscess(s);
  5. anatomical bronchial obstruction;
  6. suspected atypical pneumonia;
  7. chemical pneumonitis (e.g., inhalation injury);
  8. cystic fibrosis
* Immunocompromised patients, including those with neutropenia NOT due to the current infection (absolute neutrophil count < 500/mm3), leukemia, lymphoma, human immunodeficiency virus (HIV) infection with CD4 count < 200 cells/mm3, or splenectomy; those who are early post-transplantation (< 3 months post-transplant, or > 3 months post-transplant with evidence of organ rejection by clinical criteria, pathologic confirmation, or modification of immunosuppression within the past 4 weeks), are on cytotoxic chemotherapy, or are on high-dose steroids (e.g., > 40 mg of prednisone or its equivalent [> 160 mg hydrocortisone, > 32 mg methylprednisolone, > 6 mg dexamethasone, > 200 mg cortisone] daily for > 2 weeks)
* Evidence of significant renal impairment (serum creatinine > 4.0 mg/dL within 24 hours prior to screening). If serum creatinine is >2.0 mg/dL, site must be capable of performing continuous renal replacement therapy, if clinically indicated. Patients with serum creatinine > 4.0 mg/dL and being treated with continuous renal replacement therapy (continuous venous-venous hemofiltration or continuous venous-venous hemodialysis) or chronic hemodialysis are eligible
* Evidence of ototoxicity (history of hearing aid use prior to current hospitalization)
* Evidence of hepatotoxicity (alanine aminotransferase [ALT] or aspartate aminotransferase [AST] >3X the upper limit of normal value within 24 hours prior to screening)
* Positive urine and/or serum beta-hCG pregnancy test (only in women of reproductive age)
* On mechanical ventilation for > 28 days
* Glasgow Coma Scale score =3 at Screening
* Participating in or has participated in other investigational interventional studies (drug or device) within the last 30 days (or 5 times the half-life of the previously administered investigational compound, whichever is longer) prior to study treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2013-12; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marin Kollef, M.D., Principal Investigator — Washington University School of Medicine
Locations (35):
- United States (16):
  - Los Angeles, California
  - Gainesville, Florida
  - Jacksonville, Florida
  - Chicago, Illinois
  - Hazard, Kentucky
  - Lexington, Kentucky
  - Boston, Massachusetts
  - Burlington, Massachusetts
  - Springfield, Massachusetts
  - Detroit, Michigan
  - St Louis, Missouri
  - Omaha, Nebraska
  - Oklahoma City, Oklahoma
  - Knoxville, Tennessee
  - El Paso, Texas
  - Houston, Texas
- France (5):
  - Limoges, Limousin
  - Orléans, Loiret
  - Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - Tours
  - Colombes, Île-de-France Region
- Greece (4):
  - Alexandroupoli, Evros
  - Athens
  - Ioannina
  - Larissa
- Hungary (2):
  - Debrecen, Hajdú-Bihar
  - Budapest
- San Juan, Puerto Rico
- Spain (3):
  - Palma de Majorca, Balearic Islands
  - Getafe, Madrid
  - Barcelona
- Turkey (Türkiye) (4):
  - Ankara, Ankara
  - Ankara
  - Istanbul
  - Trabzon

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kollef MH, Ricard JD, Roux D, Francois B, Ischaki E, Rozgonyi Z, Boulain T, Ivanyi Z, Janos G, Garot D, Koura F, Zakynthinos E, Dimopoulos G, Torres A, Danker W, Montgomery AB. A Randomized Trial of the Amikacin Fosfomycin Inhalation System for the Adjunctive Therapy of Gram-Negative Ventilator-Associated Pneumonia: IASIS Trial. Chest. 2017 Jun;151(6):1239-1246. doi: 10.1016/j.chest.2016.11.026. Epub 2016 Nov 24. PMID 27890714
- See also: MedlinePlus related topics: Antibiotics — http://www.nlm.nih.gov/medlineplus/antibiotics.html
- See also: MedlinePlus related topics: Pneumonia — http://www.nlm.nih.gov/medlineplus/pneumonia.html
- See also: Drug Information available for amikacin — http://druginfo.nlm.nih.gov/drugportal/ProxyServlet?mergeData=true&objectHandle=DBMaint&APPLICATION_NAME=drugportal&actionHandle=default&nextPage=jsp/drugportal/ResultScreen.jsp&TXTSUPERLISTID=0037517285&QV1=AMIKACIN
- See also: Drug information available for fosfomycin — http://druginfo.nlm.nih.gov/drugportal/ProxyServlet?mergeData=true&objectHandle=DBMaint&APPLICATION_NAME=drugportal&actionHandle=default&nextPage=jsp/drugportal/ResultScreen.jsp&TXTSUPERLISTID=0023155024&QV1=FOSFOMYCIN
- See also: U.S. FDA Resources — http://www.clinicaltrials.gov/ct2/info/fdalinks

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The trial was designed to have 150 patients, hoping to have at least 140 patients with proven gram negative pneumonia. The trial was terminated at 143 when that goal was achieved.
Period: Overall Study
Arm/Group | Amikacin Fosfomycin Inhalation Solution | Aerosolized Placebo
Started | 71 | 72
Completed | 54 | 58
Not Completed | 17 | 14
Not completed — Adverse Event | 0 | 1
Not completed — Death | 16 | 11
Not completed — Lost to Follow-up | 0 | 2
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Amikacin Fosfomycin Inhalation Solution | Aerosolized Placebo | Total
Number analyzed (Participants) | 71 | 72 | 143
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 36 | 29 | 65
  >=65 years | 35 | 43 | 78
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 25 | 44
  Male | 52 | 47 | 99
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 41 | 41 | 82
  Unknown or Not Reported | 28 | 29 | 57
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 43 | 43 | 86
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 22 | 24 | 46
Region of Enrollment [Number; unit: participants]
  United States | 13 | 19 | 32
  Europe | 58 | 53 | 111

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Clinical Pulmonary Infection Score (CPIS) For Each Patient, Value Obtained From a Daily Assessment Over the 10 Day Study Period Was Compared to Baseline, and the LSM Data Represent the Change From Baseline Data Over All Days .
Description: Change from baseline in Clinical Pulmonary Infection Score (CPIS) For each patient, value obtained from a daily assessment over the 10 day study period was compared to baseline, and the LSM data represent the change from baseline data over all days. Daily CPIS will be determined by one blinded, central reviewer in order to minimize inter-observer variability. The scale ranges from 0 to 13, with 13 being the worst. The value of zero would be a healthy patient with no evidence of pneumonia. For each patient, there was a daily assessment for the 10 day study period.
Time Frame: 10 day treatment period.
Population: MITT
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Amikacin Fosfomycin Inhalation Solution | Aerosolized Placebo
Number analyzed (Participants) | 71 | 71
units on a scale | -0.76 (0.403) | -0.88 (0.391)

2. Secondary Outcome: Composite Endpoint of Mortality and Clinical Cure
Description: The hierarchical composite endpoint of mortality, then clinical cure (defined as both absence of Gram-negative bacteria and CPIS at Day 14 < 6). The tables reflect a winner of matched pairs, ties are not noted.
Time Frame: Day 1 - Day 28
Population: MITT
Measure: Number; unit: participants
Arm/Group | Amikacin Fosfomycin Inhalation Solution | Aerosolized Placebo
Number analyzed (Participants) | 71 | 71
participants
  Mortality first | 10 | 10
  Clinical Cure first | 15 | 18

3. Secondary Outcome: Composite Endpoint of Mortality and Ventilator-free Days
Description: The hierarchical composite endpoint of mortality, then ventilator-free days. The table reflects winners of matched pairs, ties are not noted.
Time Frame: Day 1- Day 28
Population: MITT
Measure: Number; unit: participants
Arm/Group | Amikacin Fosfomycin Inhalation Solution | Aerosolized Placebo
Number analyzed (Participants) | 71 | 71
participants
  Mortality first | 10 | 10
  Ventilator free days | 13 | 27

4. Secondary Outcome: Number of Days Free of Mechanical Ventilation From Day 1 Through Day 28
Description: Number of days free of mechanical ventilation from Day 1 through Day 28 mean days.
Time Frame: Day 1 - Day 28
Population: MITT
Measure: Mean (Standard Deviation); unit: Days ± SD
Arm/Group | Amikacin Fosfomycin Inhalation Solution | Aerosolized Placebo
Number analyzed (Participants) | 71 | 71
Days ± SD | 9.8 (9.71) | 12.5 (9.72)

5. Secondary Outcome: Number of ICU Days From Day 1 Through Day 28
Time Frame: Day 1 - Day 28
Population: MITT
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Amikacin Fosfomycin Inhalation Solution | Aerosolized Placebo
Number analyzed (Participants) | 71 | 71
Days | 28.9 (12.44) | 26.2 (12.44)

6. Secondary Outcome: Microbiological Response Rates in Patients Positive for Multi-drug Resistant Gram-negative Bacteria
Description: Microbiological response rates at Day 14 in patients whose pre-study treatment bronchoalveolar lavage (BAL) was positive for multi-drug resistant Gram-negative bacteria. Response is defined as not have a positive tracheal aspirate culture on Day 14
Time Frame: Day 14
Population: patients with MDR bacteria at baseline BAL
Measure: Count of Participants; unit: Participants
Arm/Group | Amikacin Fosfomycin Inhalation Solution | Aerosolized Placebo
Number analyzed (Participants) | 23 | 16
Participants | 10 | 7

7. Secondary Outcome: Mortality From Day 1 Through Day 28
Description: Mortality from Day 1 through Day 28, all causes, does not reflect just infection only
Time Frame: Day 1 - Day 28
Population: MITT
Measure: Number; unit: participants
Arm/Group | Amikacin Fosfomycin Inhalation Solution | Aerosolized Placebo
Number analyzed (Participants) | 71 | 71
participants | 17 | 12

8. Secondary Outcome: Clinical Relapse Rate
Description: Clinical relapse rates (defined as a new episode of pneumonia requiring reinstitution of IV antibiotics) from Day 11 through Day 28
Time Frame: Day 11 - Day 28
Population: MITT
Measure: Number; unit: participants
Arm/Group | Amikacin Fosfomycin Inhalation Solution | Aerosolized Placebo
Number analyzed (Participants) | 71 | 71
participants | 10 | 14

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Amikacin Fosfomycin Inhalation Solution | Aerosolized Placebo
Serious Adverse Events (participants affected / at risk) | 28/71 | 27/72
Other Adverse Events (participants affected / at risk) | 54/71 | 58/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amikacin Fosfomycin Inhalation Solution (N=71) | Aerosolized Placebo (N=72)
Septic shock (Infections and infestations) | 4 (4) | 6 (6)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (5)
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 2 (2)
Pneumonia (new pathogen than baseline) (Infections and infestations) | 1 (1) | 2 (2)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cardiac arrest (Cardiac disorders) | 2 (2) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 1 (1)
Lung abscess (Infections and infestations) | 0 (0) | 1 (1)
Meningitis (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Pseudomonal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Systemic candida (Infections and infestations) | 0 (0) | 1 (1)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amikacin Fosfomycin Inhalation Solution (N=71) | Aerosolized Placebo (N=72)
Hyopokalaemia (Metabolism and nutrition disorders) | 6 (6) | 6 (8)
Septic shock (Infections and infestations) | 4 (4) | 7 (7)
Pneumonia (Infections and infestations) | 5 (5) | 5 (5)
Sepsis (Infections and infestations) | 5 (5) | 4 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 5 (6)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 2 (2)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (6) | 1 (1)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 4 (5)
Nausea (Gastrointestinal disorders) | 1 (1) | 5 (5)
Constipation (Gastrointestinal disorders) | 2 (3) | 3 (3)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No